CLINICAL TRIAL: NCT07397234
Title: Thyroid Cartilage Plane Versus Superior Laryngeal Nerve Space for Ultrasound-guided Superior Laryngeal Nerve Block in Awake Tracheal Intubation: a Randomised Non-inferiority Clinical Trial
Brief Title: Thyroid Cartilage Plane VS Superior Laryngeal Nerve Space Block in Awake Tracheal Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Tao Shan, Attending physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: KY20260108-04
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Superior Laryngeal Nerve Block
Keywords: Thyroid Cartilage plane; Superior laryngeal nerve space; Difficult airway; Superior Laryngeal Nerve; Awake tracheal intubation; Nerve block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superior Laryngeal Nerve Space Block Group (C Group) (Active Comparator): All patients received topical oral and pharyngeal anesthesia using 2.4% lidocaine spray. The pharyngeal surface was sprayed twice, with each spray lasting one second, and repeated after a 5-minute interval. Under ultrasound guidance, the needle was advanced step by step into the potential space between the relevant muscle groups and the thyrohyoid membrane. When the needle tip contacted the surface of the thyrohyoid membrane and slightly penetrated the submembranous tissue, negative aspiration was confirmed, and 2.5 mL of 2% lidocaine was injected into the space on each side. Subsequently, performing fiberoptic bronchoscope-guided subglottis and tracheal surface topical anesthesia using 5ml of 2% lidocaine. After completing surface anesthesia, performing fiberoptic bronchoscope-guided tracheal intubation.
  Interventions: Procedure: Ultrasound-guided bilateral Superior Laryngeal Nerve Space Block
- Thyroid Cartilage Plane Block Group (T Group) (Experimental): All patients received topical oral and pharyngeal anesthesia using 2.4% lidocaine spray. The pharyngeal surface was sprayed twice, with each spray lasting one second, and repeated after a 5-minute interval. Ultrasound-guided bilateral Thyroid Cartilage Plane Block is performed using the thyroid cartilage as an anatomical landmark. 2.5ml of 2% lidocaine is injected on the surface of the thyroid cartilage each side. Subsequently, performing fiberoptic bronchoscope-guided subglottis and tracheal surface topical anesthesia using 2% lidocaine 5ml. After completing surface anesthesia, performing fiberoptic bronchoscope-guided tracheal intubation.
  Interventions: Procedure: Ultrasound-guided bilateral Thyroid Cartilage Plane Block

INTERVENTIONS:
Procedure: Ultrasound-guided bilateral Thyroid Cartilage Plane Block — Use a SonoSite high-frequency linear array transducer (5-13 MHz, SonoSite, USA). Placing the transducer parallel to the spine on one side of the neck, ensuring clear visualization of the thyroid cartilage under ultrasound. Using the out-of-plane technique to visualize the needle insertion path and tip. Once the needle tip contacts the cranial half of the thyroid cartilage, injecting 2.5ml of 2% lidocaine on the surface of the thyroid cartilage each side.
  Arms: Thyroid Cartilage Plane Block Group (T Group)
Procedure: Ultrasound-guided bilateral Superior Laryngeal Nerve Space Block — Use a SonoSite high-frequency linear array transducer (5-13 MHz, SonoSite, USA). Placing the transducer parallel to the spine on one side of the neck, ensuring clear visualization of the superior laryngeal nerve space under ultrasound. Using the out-of-plane technique to visualize the needle insertion path and tip. 2% lidocaine 2.5ml was injected into the space between the thyrohyoid membrane and muscle groups above.
  Arms: Superior Laryngeal Nerve Space Block Group (C Group)

SUMMARY:
The aim of this clinical trial is to compare the effectiveness and safety of ultrasound-guided thyroid cartilage plane approach with the superior laryngeal nerve space approach for superior laryngeal nerve block in awake tracheal intubation. Patients were randomized into the thyroid cartilage plane block group (T group) or the superior laryngeal nerve space block group (C group). In Group T, bilateral thyroid cartilage plane block was performed under ultrasound with thyroid cartilage as the landmark, and local anesthetic was injected on the surface of the thyroid cartilage. In Group C, local anesthetic was injected into the space between the thyrohyoid membrane and muscle groups above.

We aim to evaluate whether the thyroid cartilage plane approach is not inferior to the superior laryngeal nerve space approach for ultrasound-guided superior laryngeal nerve block in awake tracheal intubation

DETAILED DESCRIPTION:
After entering the operation room, ECG, SPO2, and invasive blood pressure were monitored. Sedation was facilitated. The proper anaesthesia depth was maintained at 60-80 using the bispectral index. Additionally, 0.5 mg of Penehyclidine Hydrochloride was injected intravenously once the venous access was established. 100% oxygen 4 L min-1 was administered with a nasal cannula throughout the procedure. All patients received topical pharyngeal anesthesia using lidocaine spray. We used a 5-12 MHz linear probeto perform bilateral block. The probe was placed parasagittally to locate the thyroid cartilage and superior laryngeal nerve space. After identification of related structure, we advanced a 22-gauge needle medial to the transducer at the upper half of the thyroid cartilage laminae until it touched the laminae or superior laryngeal nerve space using the out-of-plane technique. The correct location of the needle tip in the fascial deep to the muscle groups was confirmed by injecting 0.5-1 ml saline. A total of 2% lidocaine 2.5 ml was administered after negative aspiration bilaterally. "Spray-as-you-go" technique guided by a fiberoptic bronchoscope was performed to the tracheal with 5 ml of 2% lidocaine. After airway anesthesia, intubation completed.

The primary outcome was the proportion of acceptable intubation conditions (AIC). Secondary outcomes were the performance time, Ramsay sedation score, the patient's cough condition, comfort score, and tracheal tube tolerance score and other perioperative complications including airway hemorrhage and superior laryngeal nerve damage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for awake tracheal intubation under general anesthesia.
2. Patients with difficult airways (e.g., limited cervical spine mobility, full stomach, partial airway obstruction, craniofacial deformities or trauma, micrognathia, mouth opening <3cm, Mallampati III or IV classification) posing challenges for mask ventilation or intubation.
3. Age between 18 and 85 years old.
4. Gender is not restricted.
5. ASA classification of I - III.

Exclusion Criteria:

1. Cardiovascular dysfunction or arterial aneurysms.
2. Mental or neurological disorders or concomitant arterial aneurysms.
3. Infection at the puncture site.
4. Allergy to local anesthetics.
5. Continuous use of antiplatelet or anticoagulant medications preoperatively.
6. Hoarseness or coughing while drinking water.
7. Bronchial asthma.
8. Participation in other clinical trials within the previous 3 months before enrollment 9.r current participation in other clinical trials.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with acceptable intubation conditions (AIC) | Upon intubation
  The evaluation of the intubation condition was based on the Cormack-Lehane classification, vocal cord movement, 5-point reaction scale, and severity of coughing.
  Clinically, AIC was defined when each part was scaled to Grade 1 or Grade 2. The proportion of AIC = number of participants with AIC/number of participants who received ATI in each group.

SECONDARY OUTCOMES:
Quality of airway anesthesia | Upon intubation
  The quality of airway anesthesia assessed on a 5-point scale,Quality of airwayanesthesia was graded as: 0=no coughing or gagging in response to intubation, 1=mild coughing and/or gaggingthat did not hinder intubation, 2=moderate coughing and/or gagging that interfered minimally with intubation,3=severe coughing and/or gagging that made intubation difficult and 4=very severe coughing and/or gaggingthat required additional local anesthetic and/or change in technique.The lower grade means a better quality of airway anesthesia.
Mean Arterial Pressure | T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediately after tracheal tube insertion,T3: 5 minutes after successful intubation
  Stable blood pressure indicates a good neural blockade effect.
Heart Rate | T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediately after tracheal tube insertion,T3: 5 minutes after successful intubation
  Time Frame: T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediatelyafter tracheal tube insertion,T3: 5 minutes after successful intubation
Ramsay Sedation Score | T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediately after tracheal tube insertion,T3: 5 minutes after successful intubation
  The Ramsay Sedation Score is as follows: 6 points for unarousable, 5 points for slow response to stimulus, 4points for asleep but easily aroused, 3 points for quiet and cooperative with orientation, 2 points for asleep,anxious, restless, and 1 point for asleep, agitated, and restless. Satisfactory sedation falls within 2-4 points,while oversedation is indicated by 5-6 points.
The number of patients with lowered pitch | Before intubation
  A lowered pitch might indicate a good neural blockade effect.
The time needed for blockade procedure | From ultrasounography localization to completion of local anesthetic administration
  The neural blockade procedure time reflects the ease of the operation, with a shorter time indicating a simpler neural blockade procedure.
Record coughing in patients when the fiberoptic bronchoscope touches the glottis | Before intubation
  The patient's coughing upon contact of the fiberoptic bronchoscope with the vocal cords before intubation reflects the effectiveness of neural blockade. A lower degree of coughing indicates a better neural blockadeeffect. 1 point for no response, 2 points for mild cough, 3 points for severe cough.
The tolerance score after the tube insertion | Five minutes after successful intubation
  The tolerance of the tube reflects the patient's tolerance to awake tracheal intubation. A higher level of tolerance indicates a better neural blockade effect. 3 points for severe resistance requiring immediate general anesthesia, 2 points for restlessness and mild resistance, 1 point for cooperation.
Adverse reactions such as coughing and nausea/vomiting | During intubation
  The lower the incidence of coughing, nausea, and vomiting, the better the neural blockade effect.
Occurrences of sore throat and lowered pitch | Post-extubation,24 hours after surgery
  Pharyngeal pain and decreased vocal tone are used to assess postoperative complications of neural blockade.
Total procedure time needed for awake intubation | From the initiation of topical anesthesia to the accomplishment of tracheal intubation
  The total procedure time reflects the ease of the operation, with a shorter time indicating a simpler procedure.
Airway hemorrhage or nerve damage | During intubation
  Observation of bleeding of the laryngeal mucosa via fiberoptic bronchoscope or observation of bloody secretions via coughing or suction

CONTACTS AND LOCATIONS:
Overall Officials: Tao Shan, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No